CLINICAL TRIAL: NCT03456427
Title: Patient-Assisted Compression in 3D - Impact on Image Quality and Workflow
Acronym: 3D PAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 124.03-2017-GES-0005
Record Dates: First submitted 2018-02-23; First posted 2018-03-07 (Actual); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Study Participants (Other): All subjects will undergo standard of care imaging on one breast. The other breast will be imaged using Patient-Assisted Compression (PAC), followed by Technologist-controlled (TC) Compression.
  Interventions: Device: Patient-Assisted Compression (PAC); Device: Technologist-Controlled (TC) Compression

INTERVENTIONS:
Device: Patient-Assisted Compression (PAC) — The technologist will properly position the breast and apply minimum compression. The subject will be instructed to apply compression as the technologist ensures the breast tissue is in appropriate position and tautness. The technologist will then guide the subject to achieve appropriate compression level, sufficient but not excessive, and the image will be acquired. This will be done for both standard views Craniocaudal (CC) & Mediolateral Oblique (MLO).
Device: Technologist-Controlled (TC) Compression — TC compression will be conducted per standard of care practices at the site.

SUMMARY:
Patient-assisted compression (PAC) allows the patient to participate in controlling the amount of compression force during mammography and is a personalized approach that has demonstrated successful reduction in discomfort experienced during mammography. General Electric Healthcare's Senographe Pristina, an innovative mammography platform that provides both two-dimensional (2D) and three-dimensional (3D) imaging capabilities, offers both standard and patient-assisted compression modes. This study will evaluate image quality and clinical workflow as it relates to use of PAC with the Senographe Pristina 3D.

DETAILED DESCRIPTION:
The study population will consist of adult asymptomatic women presenting for screening 2D mammography. One breast of each subject will be identified as the "breast of interest," which will undergo study-specific 3D imaging consisting of two-view (craniocaudal and mediolateral oblique) PA compression and image acquisition, followed by two-view technologist-controlled (TC) compression and image acquisition. The breast of interest will be randomly assigned to either the first breast imaged during the exam or the second breast imaged. TC compression and imaging, and procedures performed on the subject's other breast will be conducted per standard of care.

Following image acquisition, 3D image quality evaluation will be conducted by Mammography Quality Standards Act-qualified readers. Prior to the reading session, images will be de-identified and the following information will be removed from the DICOM header to blind readers to the compression mode used during acquisition: time stamp, compression force, and breast thickness. The image sets will also be randomized for presentation during the image attribute reviews. Two (2) readers will evaluate each PAC and TC compression image set collected from each subject's breast of interest and assess the acceptability of image attributes, as defined in the Guidance for Industry and FDA Staff - Class II Special Controls Guidance Document: Full-Field Digital Mammography System (2012). A third reader will provide adjudication, if there is disagreement for a given image set's overall clinical image quality.

Workflow data, including the incidence of technologist intervention during acquisition and need for repeat image acquisition, will also be collected.

The proportion of PAC image sets that are of equal or higher acceptability than TC image sets will be calculated. A 95% confidence interval will be calculated using asymptotic method with continuity correction. The proportion of image sets indicated for repeated image acquisition when using PA mode or TC mode will be summarized. Other endpoint data will be summarized using descriptive statistics. No statistical hypothesis is being tested in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Are women aged 40 years or older;
2. Are asymptomatic and scheduled for screening mammography;
3. Have left and right breasts;
4. Have breast sizes compatible with the dimensions of a 24 x 31 cm image detector, without anatomical cut-off;
5. Are documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy;
6. Are able and willing to comply with study procedures; and
7. Are able and willing to provide written informed consent to participate.

Exclusion Criteria:

1. Are women aged 40 years or older;
2. Are asymptomatic and scheduled for screening mammography;
3. Have left and right breasts;
4. Have breast sizes compatible with the dimensions of a 24 x 31 cm image detector, without anatomical cut-off;
5. Are documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy;
6. Are able and willing to comply with study procedures; and
7. Are able and willing to provide written informed consent to participate.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boca Raton Regional Hospital, Boca Raton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All subjects underwent standard of care imaging on one breast. The other breast was imaged using Patient-Assisted Compression (PAC), followed by Technologist-controlled (TC) Compression.
  Patient-Assisted Compression (PAC): The technologist properly positioned the breast and applied minimum compression. The subject was instructed to apply compression as the technologist ensures the breast tissue is in appropriate position and tautness. The technologist will then guide the subject to achieve appropriate compression level, sufficient but not excessive, and the image was acquired. This was done for both standard views CC & MLO.
  Technologist-Controlled (TC) Compression: TC compression was conducted per standard of care practices at the site.
Period: Overall Study
Arm/Group | All Study Participants
Started | 36
Completed | 33
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All subjects will undergo standard of care imaging on one breast. The other breast will be imaged using Patient-Assisted Compression (PAC), followed by Technologist-controlled (TC) Compression.
  Patient-Assisted Compression (PAC): The technologist will properly position the breast and apply minimum compression. The subject will be instructed to apply compression as the technologist ensures the breast tissue is in appropriate position and tautness. The technologist will then guide the subject to achieve appropriate compression level, sufficient but not excessive, and the image will be acquired. This will be done for both standard views CC & MLO.
  Technologist-Controlled (TC) Compression: TC compression will be conducted per standard of care practices at the site.
Arm/Group | All Study Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.45 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Menopausal Status [Count of Participants; unit: Participants]
  Post-Menopausal | 29
  Perimenopause | 2
  Pre-Menopausal | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Acceptable Overall Image Quality
Description: The primary objective is to compare the percentage of acceptable overall image quality in unilateral two-view (CC and MLO) breast images acquired using Patient-Assisted Compression and Technologist Compression modes.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Patient Assisted Compression: All subjects will undergo standard of care imaging on one breast. The other breast will be imaged using Patient-Assisted Compression (PAC), followed by Technologist-controlled (TC) Compression.
  Patient-Assisted Compression (PAC): The technologist will properly position the breast and apply minimum compression. The subject will be instructed to apply compression as the technologist ensures the breast tissue is in appropriate position and tautness. The technologist will then guide the subject to achieve appropriate compression level, sufficient but not excessive, and the image will be acquired. This will be done for both standard views CC & MLO.
- All Study Participants: Technologist Compression: All subjects will undergo standard of care imaging on one breast. The other breast will be imaged using Patient-Assisted Compression (PAC), followed by Technologist-controlled (TC) Compression.
  Technologist-Controlled (TC) Compression: TC compression will be conducted per standard of care practices at the site.
Arm/Group | All Study Participants: Patient Assisted Compression | All Study Participants: Technologist Compression
Number analyzed (Participants) | 33 | 33
Participants
  Image Quality: Acceptable | 30 | 33
  Image Quality: Unacceptable | 3 | 0

2. Secondary Outcome: Number of Repeat Image Acquisitions
Description: To evaluate the need for repeat image acquisition when using Patient-Assisted Compression and Technologist Compression modes.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants: Patient Assisted Compression | All Study Participants: Technologist Compression
Number analyzed (Participants) | 33 | 33
Participants
  Technologist-Indicated Repeat Acquisitions: Repeat Acquisitions Indicated | 1 | 0
  Technologist-Indicated Repeat Acquisitions: Repeat Acquisition not Indicated | 32 | 33
  Reader-Indicated Repeat Acquisitions: Repeat Acquisitions Indicated | 3 | 3
  Reader-Indicated Repeat Acquisitions: Repeat Acquisition not Indicated | 30 | 30

3. Secondary Outcome: Percentage of Acceptable Mammographic Attributes
Description: To evaluate the percentage of acceptable mammographic attributes for unilateral two-view breast images acquired using Patient-Assisted Compression and Technologist Compression modes.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants: Patient Assisted Compression | All Study Participants: Technologist Compression
Number analyzed (Participants) | 33 | 33
Participants
  Breast Positioning: Acceptable | 29 | 32
  Breast Positioning: Unacceptable | 4 | 1
  Exposure and Visualization: Acceptable | 33 | 33
  Exposure and Visualization: Unacceptable | 0 | 0
  Breast Compression: Acceptable | 31 | 32
  Breast Compression: Unacceptable | 2 | 1
  Sharpness due to Motion: Acceptable | 32 | 31
  Sharpness due to Motion: Unacceptable | 1 | 2
  Image Contrast: Acceptable | 33 | 33
  Image Contrast: Unacceptable | 0 | 0
  Tissue Visibility at skin line: Acceptable | 31 | 32
  Tissue Visibility at skin line: Unacceptable | 2 | 1
  Noise: Acceptable | 33 | 33
  Noise: Unacceptable | 0 | 0
  Artifacts due to image processing or other factors: Acceptable | 33 | 33
  Artifacts due to image processing or other factors: Unacceptable | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03456427/Prot_SAP_000.pdf